CLINICAL TRIAL: NCT01634724
Title: Study of Effect of GnRHa Withdrawal at Late Stage of Long Protocol on the Risk of Ovarian Hyper-stimulation in Patients With Polycystic Ovary (PCO) Undergoing in Vitro Fertilization/Intracytoplasmic Sperm Injection Cycles
Brief Title: GnRH Agonist (GnRHa) Withdrawal at Late Stage of Long Protocol and the Incidence of Ovarian Hyper-stimulation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanjing University (Other)
Responsible Party: Principal Investigator, Li-jun Ding, Associate Professor, Nanjing University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: NJGLHRMCSUN1
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Infertile High-risk Patients With Polycystic Ovaries
Keywords: GnRH agonist withdrawal; OHSS; E2; VEGF

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GnRH agonist withdrawal (Experimental): All the patients received a midluteal long GnRH agonist (GnRH-a) and a gonadotropins (recombinant FSH) stimulation protocol. When the diameter of one or more follicles was ≥ 14 mm, GnRHa (0.05mg/d) was withheld in the study group.
  Interventions: Drug: a drug withdrawal during the long protocol
- control group (No Intervention): All the patients received a midluteal long GnRH agonist (GnRH-a) and a gonadotropins (recombinant FSH) stimulation protocol. In the control group, GnRHa (triptorelin, 0.05mg/d,)was used to the day of ovulation trigger.

INTERVENTIONS:
Drug: a drug withdrawal during the long protocol — GnRHa (triptorelin,0.05mg/d) was injected stimulously with FSH before dominant follicles were ≥ 14 mm. When the diameter of one or more follicles was ≥ 14 mm, GnRHa (triptorelin,0.05mg/d) was withheld in the study group.
  Other Names: GnRH agonist wihtholding or GnRH agonist coasting
  Arms: GnRH agonist withdrawal

SUMMARY:
To test whether GnRHa withheld 2-3 days before ovulation trigger reduces the incidence of ovarian hyperstimulation syndrome (OHSS) in infertile high-risk patients with polycystic ovaries (PCOs) who have been treated with gonadotropins for in vitro fertilization (IVF) or Intracytoplasmic sperm injection (ICSI).

DETAILED DESCRIPTION:
All the patients received a midluteal long GnRH agonist (GnRH-a) and a gonadotropins (recombinant FSH) stimulation protocol. Pituitary down-regulation with GnRH agonist (triptorelin, 0.1mg/d, ×10d, then 0.05mg/d until E2 ≤40 pg/ml in serum), was initiated during the luteal phase on the cycle-day 21. Two weeks later, if E2 in serum was ≤40 pg/ml and absence of follicular activity was detected, the stimulation of ovaries was started by recombinant follicle-stimulating hormone (recFSH, Gonal-F, Serono, Switzerland) with doses ranging 150-250 IU/d. Doses were adjusted accordingly with ovarian monitoring and follicles growth. GnRHa (0.05mg/d) was injected stimulously with FSH before dominant follicles were ≥ 14 mm. When the diameter of one or more follicles was ≥ 14 mm, GnRHa (0.05mg/d) was withheld in the study group. In the control group, GnRHa was used to the day of ovulation trigger. Ovulation was induced with HCG (5000-10000 IU) when at least three follicles greater than 16mm in diameter were detected on ultrasound examination and the leading follicles reached ≥ 18 mm in diameter. Oocytes retrieval for IVF or ICSI was performed 34-36 hours later under transvaginal ultrasound guidance.

Main Outcome Measure(s): Serum E2 levels, VEGF levels in Serum and follicular fluids, retrieved oocytes, fertilization, implantation rate and pregnancy rate (PR), the rate of OHSS.

ELIGIBILITY:
Inclusion Criteria:

ninety-six infertile patients with PCOs (12 or more follicles 2-9 mm in diameter were detected in ovaries by ultrasound detection) undergoing IVF treatment were enrolled.

Exclusion Criteria:

the subjects included the followings: a basal FSH level of > 10IU/L; age >35 years; a body mass index (BMI) > 30 kg/m2; ovarian surgery radiotherapy or chemotherapy; ovarian dysfunction; endometriosis; hyperprolactinemia; thyroid dysfunction; the presence of organic pelvic diseases.

Ages: 23 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2012-07; Primary Completion 2012-07 (Actual); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
incidence of ovarian hyperstimulation | two weeks
  Ovarian hyperstimulation syndrome is a complication from some forms of fertility medication. Most cases are mild, but a small proportion are severe. Symptoms are set into 3 categories: mild, moderate, and severe.

SECONDARY OUTCOMES:
pregnancy rate in the patients with IVF or ICSI | one month

CONTACTS AND LOCATIONS:
Overall Officials: Hai-xiang Sun, ph.D, Study Director — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Research Room of Reproductive Medicine, The Outpatient Building of Drum Tower Hospital, Nanjing, Jiangsu, China

REFERENCES:
- [Background] Ho Yuen B, Nguyen TA, Cheung AP, Leung PC. Clinical and endocrine response to the withdrawal of gonadotropin-releasing hormone agonists during prolonged coasting. Fertil Steril. 2009 Aug;92(2):499-507. doi: 10.1016/j.fertnstert.2008.06.039. Epub 2008 Aug 15. PMID 18706551